CLINICAL TRIAL: NCT04735822
Title: A 2-Part, Phase I Study to Evaluate the Taste Profile of Belumosudil Oral Suspensions & Assess Relative Bioavailability of the Selected Belumosudil Oral Suspension Formulation Compared With Oral Tablets in Healthy Male Subjects
Brief Title: A Phase I Study to Evaluate the Taste of Belumosudil Oral Suspensions & Assess Relative Bioavailability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD025-111; 2020-003446-37 (EudraCT Number)
Record Dates: First submitted 2021-01-13; First posted 2021-02-03 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
Keywords: Belumosudil; KD025; SLx-2119; ROCK inhibitor; Healthy male subjects
MeSH Terms: interventions — KD025

STUDY DESIGN:
Intervention Model Description: Part 1: Single center, open-label, randomized, 6-arm design to assess the taste profile of different novel belumosudil in bottle formations in 12 healthy male subjects.
  Part 2: Single center, open-label, randomized, 3-arm, design to assess the relative bioavailability of a selected belumosudil suspension formulation compared to the oral belumosudil tablet reference and the effect of food on the selected belumosudil suspension formulation in 18 health male subjects
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1: Belumosudil Sequence ABFCED (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen A (delivered by Vehicle 1); Regimen B (delivered by Vehicle 2); Regimen F (delivered by Vehicle 6); Regimen C (delivered by Vehicle 3); Regimen E (delivered by Vehicle 5); Regimen D (delivered by Vehicle 4);
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence ABFCED
- Part 1: Belumosudil Sequence BCADFE (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen B (delivered by Vehicle 2); Regimen C (delivered by Vehicle 3); Regimen A (delivered by Vehicle 1); Regimen D (delivered by Vehicle 4); Regimen F (delivered by Vehicle 6); Regimen E (delivered by Vehicle 5)
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence BCADFE
- Part 1: Belumosudil Sequence CDBEAF (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen C (delivered by Vehicle 3); Regimen D (delivered by Vehicle 4); Regimen B (delivered by Vehicle 2); Regimen E (delivered by Vehicle 6); Regimen A (delivered by Vehicle 1); Regimen F (delivered by Vehicle 6)
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence CDBEAF
- Part 1: Belumosudil Sequence DECFBA (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen D (delivered by Vehicle 4); Regimen E (delivered by Vehicle 5); Regimen C (delivered by Vehicle 3); Regimen F (delivered by Vehicle 6); Regimen B (delivered by Vehicle 2); Regimen A (delivered by Vehicle 1)
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence DECFBA
- Part 1: Belumosudil Sequence EFDACB (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen E (delivered by Vehicle 5); Regimen F (delivered by Vehicle 6); Regimen D (delivered by Vehicle 4); Regimen A (delivered by Vehicle 1); Regimen C (delivered by Vehicle 3); Regimen B (delivered by Vehicle 2)
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence EFDACB
- Part 1: Belumosudil Sequence FAEBDC (Experimental): Subjects receive 1 dose of belumosudil 40 mg/mL in oral suspension in the following sequence: Regimen F (delivered by Vehicle 6); Regimen A (delivered by Vehicle 1); Regimen E (delivered by Vehicle 5); Regimen B (delivered by Vehicle 2); Regimen D (delivered by Vehicle 4); Regimen C (delivered by Vehicle 3).
  Interventions: Drug: Part 1: Belumosudil 40 mg/mL Sequence FAEBDC
- Part 2: Belumosudil Sequence GHI (Experimental): Subjects receive 1 dose in the following sequence; Regimen G (belumosudil 200 mg tablet fed); Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted); Regimen I (powder for oral suspension or oral suspension belumosudil 200 mg fed)
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence GHI
- Part 2: Belumosudil Sequence HIG (Experimental): Subjects receive 1 dose in the following sequence: Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted); Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fed); Regimen G (belumosudil 200 mg tablet fed)
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence HIG
- Part 2: Belumosudil Sequence IGH (Experimental): Subjects receive 1 dose in the following sequence: Regimen I (powder for oral suspension or oral suspension belumosudil 200 mg fed); Regimen G (belumosudil 200 mg tablet fed); Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted)
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence IGH
- Part 2: Belumosudil Sequence IHG (Experimental): Subjects receive 1 dose in the following sequence: Regimen I (powder for oral suspension or oral suspension belumosudil 200 mg fed); Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted); Regimen G (belumosudil 200 mg tablet fed)
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence IHG
- Part 2: Belumosudil Sequence GIH (Experimental): Subjects receive 1 dose in the following sequence: Regimen G (belumosudil 200 mg tablet fed); Regimen I (powder for oral suspension or oral suspension belumosudil 200 mg fed); Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted)
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence GIH
- Part 2: Belumosudil Sequence HGI (Experimental): Subjects receive 1 dose in the following sequence: Regimen H (powder for oral suspension or oral suspension belumosudil 200 mg fasted); Regimen G (belumosudil 200 mg tablet); Regimen I (powder for oral suspension or oral suspension belumosudil 200 mg fed);
  Interventions: Drug: Part 2: Belumosudil 200 mg Sequence HGI

INTERVENTIONS:
Drug: Part 1: Belumosudil 40 mg/mL Sequence ABFCED — Oral suspension belumosudil 40 mg/mL in sequence Regimen A, then Regimen B, then Regimen F, then Regimen C, then Regimen E, then Regimen D
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence ABFCED
Drug: Part 1: Belumosudil 40 mg/mL Sequence BCADFE — Oral suspension belumosudil 40 mg/mL in sequence Regimen B, then Regimen C, then Regimen A, then Regimen D, then Regimen F, then Regimen E
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence BCADFE
Drug: Part 1: Belumosudil 40 mg/mL Sequence CDBEAF — Oral suspension belumosudil 40 mg/mL in sequence Regimen C, then Regimen D, then Regimen B, then Regimen E, then Regimen A, then Regimen F
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence CDBEAF
Drug: Part 1: Belumosudil 40 mg/mL Sequence DECFBA — Oral suspension of belumosudil 40 mg/mL in sequence Regimen D, then Regimen E, then Regimen C, then Regimen F, then Regimen B, then Regimen A
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence DECFBA
Drug: Part 1: Belumosudil 40 mg/mL Sequence EFDACB — Oral suspension of belumosudil 40 mg/mL in sequence Regimen E, then Regimen F, then Regimen D, then Regimen A, then Regimen C, then Regimen C
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence EFDACB
Drug: Part 1: Belumosudil 40 mg/mL Sequence FAEBDC — Oral suspension of belumosudil 40 mg/mL in sequence Regimen F, then Regimen A, then Regimen E, then Regimen B, then Regimen D, then Regimen C
  Other Names: KD025
  Arms: Part 1: Belumosudil Sequence FAEBDC
Drug: Part 2: Belumosudil 200 mg Sequence GHI — 1 dose of belumosudil 200 mg in sequence Regimen G (tablet), then Regimen H (oral suspension; subject fasted), then Regimen I (oral suspension; subject fed)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence GHI
Drug: Part 2: Belumosudil 200 mg Sequence HIG — 1 dose of belumosudil 200 mg in sequence Regimen H (oral suspension; subject fasted), then Regimen I (oral suspension; subject fed), then Regimen G (tablet)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence HIG
Drug: Part 2: Belumosudil 200 mg Sequence IGH — 1 dose of belumosudil 200 mg in sequence Regimen I (oral suspension; subject fed), then Regimen G (tablet), then Regimen H (oral suspension, subject fasted)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence IGH
Drug: Part 2: Belumosudil 200 mg Sequence IHG — 1 dose of belumosudil 200 mg in sequence Regimen I (oral suspension; subject fed), then Regimen H (oral suspension; subject fasted), then Regimen G (tablet)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence IHG
Drug: Part 2: Belumosudil 200 mg Sequence GIH — 1 dose of belumosudil 200 mg in sequence Regimen G (tablet), then Regimen I (oral suspension; subject fed), then Regimen H (oral suspension; subject fasted)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence GIH
Drug: Part 2: Belumosudil 200 mg Sequence HGI — 1 dose of belumosudil 200 mg in sequence Regimen H (oral suspension; subject fasted), then Regimen G (tablet), then Regimen I (oral suspension; subject fed)
  Other Names: KD025
  Arms: Part 2: Belumosudil Sequence HGI

SUMMARY:
This is a single-center, randomized, open-label, 2-part study in healthy male subjects to evaluate the taste profile of different belumosudil oral suspensions and the relative bioavailability of those chosen oral suspensions of belumosudil compared to oral tablets of belumosudil.

Part 1 is an open-label, randomized single-period study of oral suspensions of belumosudil 40 mg/mL delivered in 6 different vehicles. Approximately 12 healthy male subjects, 2 subjects in each of 6 groups, will be administered a single dose of belumosudil 40 mg/mL in 6 different vehicles (Vehicles 1, 2, 3, 4, 5, and 6) in corresponding Regimens A, B, C, D, E, and F in different sequences of the 6 vehicles. All subjects will receive 1 dose of all belumosudil in all 6 vehicles which are as follows: ABFCED; BCADFE; CDBEAF; DECFBA; EFDACB; and FAEBDC.

Part 2 is a single-center, open-label, randomized, 3-period design to assess the relative bioavailability of a selected belumosudil suspension formulation compared to the oral belumosudil. Tablet reference and the effect of food on the selected belumosudil suspension formulation in 18 healthy male subjects. Subjects will be randomized prior to the administration of the first dose of IMP to 1 of 6 treatment sequences (GHI, HIG, IGH, IHG, GIH and HGI), with 3 subjects assigned to each treatment sequence where:

Regimen G--oral belumosudil 200 mg tablet (reference) with the subject fed; Regimen H--belumosudil powder 200 mg for oral suspension or belumosudil 200 mg oral suspension with the subject fasting; and Regimen I--belumosudil 200 mg powder for oral suspension or belumosudil 200 mg oral suspension with the subject fed.

DETAILED DESCRIPTION:
PART 1

This is a single center, open-label, randomized, single period design to assess the taste profile of different novel regimens from bottles containing 1200 mg of belumosudil. Twelve healthy subjects will receive single doses of the 6 bottled oral formulations:

Regimen A: belumosudil 40 mg/mL delivered by Vehicle 1 (sterile water for irrigation); Regimen B: belumosudil 40 mg/mL delivered by Vehicle 2 (low sucralose solution); Regimen C: belumosudil 40 mg/mL delivered by Vehicle 3 (high sucralose solution); Regimen D: belumosudil 40 mg/mL delivered by Vehicle 4 (orange flavor with low sucralose solution); Regimen E: belumosudil 40 mg/mL delivered by Vehicle 5 (tropical fruit blend with low sucralose solution); Regimen F: belumosudil 40 mg/mL delivered by Vehicle 6 (lemon flavor with low sucralose solution)

Subjects will sip the belumosudil oral suspension and then spit it out. The maximum dose is belumosudil 200 mg.

On Day 1, two subjects each will be randomized to 1 of 6 treatment sequences with belumosudil:

ABFCED (2 subjects); BCADFE (2 subjects); CDBEAF (2 subjects); DECFBA (2 subjects); EFDACB (2 subjects); FAEBDC (2 subjects)

Subjects will undergo preliminary screening procedures to determine their eligibility for Part 1 of the study at a screening visit (Day -28 to Day -2 of Part 1). Subjects will be admitted to the clinical unit on the morning prior to investigational medicinal product (IMP) administration (Day -1) for confirmation of eligibility and baseline procedures. Prior to the first administration of IMP (either Day -1 or prior to the completion of breakfast [pre-dose] on Day 1), subjects will be given a training questionnaire using an example fluid (e.g., orange juice/squash).

In the evening of Day -1, subjects will receive a light snack and will then fast from all food and drink (except water). Following the overnight fast (approximately 8 hours), subjects will consume a standard breakfast. Following breakfast, subjects will brush their teeth using tap water (toothpaste will not be permitted). The first dose of IMP will be administered approximately 2 hours after breakfast has been completed.

Subjects will receive the test belumosudil from bottles in regimens according to a randomization schedule. Each regimen will follow the same study design. Subjects will receive a single dose of belumosudil 40 mg/mL as an oral suspension, which will be held in the mouth for approximately 1 minute before it is expectorated, and will subsequently complete a written taste/palatability questionnaire individually and privately. No belumosudil is to be consumed.

There will be a washout period of 30 min ± 10 min (minimum 20 min) between tasting each regimen (inclusive of palate cleansing). During this time, subjects will cleanse their palates using tap water (administered freely in 50 mL aliquots) and unsalted crackers before further tasting. It is expected that all regimens will be tasted on the same day.

A single plasma pharmacokinetic (PK) sample will be taken approximately 1 hour post-final dose (prior to discharge from the clinical unit). This sample will be retained and only analyzed in case of accidental swallowing of the formulation by a subject and/or for the purpose of investigating a possible treatment-emergent adverse event (TEAE) related to the IMP.

Subjects will remain on site until 1 hour post-final taste/palatability assessment. To ensure the ongoing well-being of the subjects, a follow-up phone call will take place 3 to 7 days after the final dose. If a subject reports any adverse events (AEs) after discharge which is a cause for concern, they will be required to attend the clinical unit for a follow-up assessment. This follow-up visit will be considered an unscheduled visit.

Following the completion of Part 1, an interim data review will be performed during which the taste/palatability assessment data will be reviewed to determine the flavor system that will be incorporated into the IMP formulation for administration in Part 2.

PART 2

This is a single-center, open-label, randomized, 3-period design to assess the relative bioavailability of a selected belumosudil suspension formulation from Part 1 compared to the belumosudil oral tablet. Eighteen subjects will receive single doses of the following:

Regimen G = 200 mg belumosudil tablet (reference drug) orally when subjects are fed; Regimen H = 200 mg belumosudil powder for oral suspension or belumosudil oral suspension when subjects are fasting; and Regimen I = 200 mg belumosudil powder for oral suspension or belumosudil oral suspension when subjects are fed.

On Day 1, three subjects each will be randomized to 1 of 6 treatment sequences with belumosudil:

GHI (3 subjects); HIG (3 subjects); IGH (3 subjects); IHG (3 subjects); GIH (3 subjects); HGI (3 subjects)

Subjects will undergo preliminary screening procedures to determine their eligibility for Part 2 of the study at a screening visit (Day -28 to Day -2 of Part 2). Subjects who have taken part in Part 1 of the study are permitted to take part in Part 2.

Each study period will follow a similar design. Subjects will be admitted to the clinical unit on the morning prior to the first IMP administration (Day -1 of Period 1) for confirmation of eligibility and baseline procedures. For Regimen H only, subjects will be given a training questionnaire using an example fluid (e.g., orange juice/squash) prior to IMP administration. This will be performed either on Day -1 (only applicable if Regimen H is administered in Period 2 or 3) or prior to the completion of breakfast (pre-dose) on Day 1.

Subjects will receive a single dose of IMP in the morning of Day 1 following an overnight fast of a minimum of 10 hours (Regimen H, fasted state) or following a standard breakfast (Regimens G and I, fed state). Blood samples will be collected at regular intervals for PK analysis. Following administration of Regimen H, subjects will complete a written taste/palatability questionnaire individually and privately.

Subjects will reside in the clinical unit for 10 consecutive nights that will cover all 3 treatment periods. All subjects will remain on site until 72 h post-final dose for safety and PK assessments. There will be a minimum washout period of 3 days between each IMP administration. To ensure the ongoing well-being of the subjects, a follow-up phone call will take place 3 to 7 days after the final dose. If a subject reports any AEs after discharge which is a cause for concern, they will be required to attend the clinical unit for a follow-up assessment. This follow-up visit will be considered an unscheduled visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 18 to 55 years inclusive at the time of signing informed consent.
3. Body mass index of 18.0 to 32.0 kg/m^2 at screening
4. Body weight ≥ 50 kg at screening
5. Must be willing and able to communicate and participate in the entire study
6. Must provide written informed consent
7. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who have received any IMP in a previous clinical research study within the 90 days prior to Day 1 (Part 2 only)
2. Subjects who are or are immediate family members of a study site or sponsor employee
3. Subjects who have previously been administered IMP in Part 2 of this study. Subjects who have taken part in Part 1 are permitted to take part in Part 2
4. Evidence of current SARS-CoV-2 infection
5. Clinically significant history or presence of acute or chronic bacterial, fungal, or viral infection (e.g., pneumonia, septicemia) within the 3 months or 90 days prior to screening
6. Any subject with clinically significant symptoms of COVID-19 in the last 4 weeks, including but not limited to fever, new and persistent cough, breathlessness or loss of taste or smell, as per the judgement of the investigator
7. Known or suspected malignancy, autoimmune disorder, or any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status or any factor that would predispose participants to develop infection (e.g., open skin lesions, recurrent issues related to poor dentition, perianal fissures, history of splenectomy, primary immunodeficiency)
8. History of any drug or alcohol abuse in the past 2 years
9. Regular alcohol consumption in males > 21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirits, 1.5 to 2 units = 125 mL glass of wine, depending on type)
10. A confirmed positive alcohol breath test at screening or admission
11. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
12. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
13. Subjects with pregnant or lactating partners
14. Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the investigator or delegate at screening
15. Clinically significant abnormal clinical chemistry, hematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are allowed.
16. Confirmed positive drugs of abuse test result.
17. Positive hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antibody results
18. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of < 80 mL/min using the Cockcroft-Gault equation (Part 2 only)
19. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory, gastrointestinal (GI) disease, or neurological or psychiatric disorder as judged by the investigator
20. Subject has a history or presence of any of the following (Part 2 only):

    * Cytopenias
    * Active GI disease requiring therapy
    * Hepatic disease and/or alanine aminotransferase or aspartate aminotransferase > upper limit of normal (ULN)
    * Renal disease and/or serum creatinine > ULN
    * Other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
21. Subjects with a history of cholecystectomy or gall stones (Part 2 only)
22. Subject has QTcF intervals >450 msec at screening or admission (Part 2 only)
23. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
24. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
25. Donation of blood or plasma within the previous 3 months or loss > 400 mL of blood
26. Subjects who are taking or have taken any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days prior to IMP administration, including proton pump inhibitors. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
27. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Taste/Palatability Questionnaire for Regimens B, C, D, E, F vs. Regimen A (Part 1 Only) | Immediately after dosing
  Comparison of Taste/Palabability Questionnaire results of (1) Regimen B (belumosudil 400 mg/mL using Vehicle 2) vs. Regimen A (belumosudil 400 mg/mL using Vehicle 1); (2) Regimen C (belumosudil 400 mg/mL using Vehicle 3) vs. Regimen A; (3) Regimen D (belumosudil 40 mg/mL using Vehicle 4) vs. Regimen A; (4) Regimen E (belumosudil 40 mg/mL using Vehicle 5) vs. Regimen A; and (5) Regimen F (belumosudil 40 mg/mL using Vehicle 5) vs. Regimen A.
  The Taste/Probability Questionnaire assess smell, sweetness, bitterness, flavor, mouth feel/texture, grittiness, and aftertaste. Subjects rate each sense on a categorical scale ranging from extreme dislike to extreme like.
Selection of Belumosudil Suspension Formulation for Part 2 | After administration of belumosudil 40 mg/mL with each of the 6 vehicles in the sequence assigned
  Selection of the belumosudil suspension formulation to be used in Part 2 of the study

SECONDARY OUTCOMES:
Pharmacokinetics (Part 2 Only): Relative Bioavailability of Regimen I vs. Regimen G | Up to 72 hours post-dose
  Comparison of Regimen I (powder for oral suspension or oral suspension of belumosudil 200 mg fed) vs. Regimen G (belumosudil 200 mg tablet fed)
Pharmacokinetics (Part 2 Only): Determination of Tlag of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the time prior to the first measurable concentration (Tlag) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of Tmax of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the time of maximum observed concentration (Tmax) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of Cmax of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the maximum observed concentration (Cmax) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of AUC(0-24) of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the area under the concentration-time curve from time 0 to 24 hours post-dose (AUC[0-24]) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of AUC(0-last) of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the area under the concentration-time curve from time 0 to the time of last measurable concentration (AUC[0-last]) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of AUC(0-inf) of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the area under the concentration-time curve from time 0 extrapolated to infinity (AUC[0-inf]) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of AUC%extrap of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the area under the concentration-time curve from the time of the last measurable concentration to infinity as a percentage of the area under the concentration-time curve extrapolated to infinity (AUC%extrap) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of t1/2 of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the terminal elimination half-life (t1/2) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of Lambda-z of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve (Lambda-z) of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of CL/F of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (belumosudil only), i.e., CL/F
Pharmacokinetics (Part 2 Only): Determination of Vz/F of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where the fraction of dose bioavailable (F) is unknown (belumosudil only), i.e., Vz/F
Pharmacokinetics (Part 2 Only): Determination of Frel Cmax of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the relative bioavailability based on Cmax, i.e., Frel Cmax, of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of Frel AUC(0-last) of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the relative bioavailability based on AUC(0-last), i.e., Frel AUC(0-last), of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): Determination of Frel AUC(0-inf) of Belumosudil 200 mg | Up to 72 hours post-dose
  Assessment of the relative bioavailability based on AUC(0-inf), i.e., Frel AUC(0-inf), of oral belumosudil 200 mg
Pharmacokinetics (Part 2 Only): MPR Cmax of Belumosudil 200 mg | Up to 72 hours post-dose
  Metabolite-to-parent ratio (MPR) based on the Cmax of metabolite KD025m1 and metabolite KD025m2 of belumosudil 200 mg orally
Pharmacokinetics (Part 2 Only): MPR AUC(0-last) of Belumosudil 200 mg | Up to 72 hours post-dose
  Metabolite-to-parent ratio (MR) based on AUC(0-last) of metabolite KD025m1 and metabolite KD025m2 only, i.e., MPR AUC(0-last)
Pharmacokinetics (Part 2 Only): MPR AUC(0-inf) of Belumosudil 200 mg | Up to 72 hours post-dose
  Metabolite-to-parent ratio based on AUC(0-inf) of metabolite KD025m1 and metabolite KD025m2, i.e., MPR AUC(0-inf)
Safety: Incidence, Intensity, and Relationship of AEs to Belumosudil 200 mg | Up to 7 days after the last dose (duration of study)
  Proportion of subjects with adverse events (AEs) overall, by intensity, and by relationship to oral belumosudil 200 mg
Safety: Incidence, Intensity, and Relationship of SAEs to Belumosudil 200 mg | Up to 7 days after the last dose (duration of study)
  Proportion of subjects with serious adverse events (SAEs) overall, by intensity, and by relationship to oral belumosudil 200 mg
Safety: Incidence, Intensity, and Relationship of AEs Leading to Discontinuation from the Study | Up to 7 days after the last dose (duration of study)
  Proportion of subjects who had AEs leading to discontinuation from the study, by intensity, and by relationship to oral belumosudil 200 mg

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, BSc, MD, DPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, England, United Kingdom